CLINICAL TRIAL: NCT07305181
Title: Screening and Identifying Abnormal Haemoglobin Fractions in a Metropolitan Area in Chattogram
Brief Title: Prevalence of Abnormal Haemoglobin Variants in Metropolitan Chattogram, Bangladesh
Acronym: Hb Variants
Status: Completed | Type: Observational
Sponsor: Bangladesh Bioscience Research Group (Network)
Collaborators: Chattogram International Dental College (Other); Chittagong Medical College and Hospital (Other); Bangladesh Medical University (Other)
Responsible Party: Principal Investigator, Pair Ahmed Jiko, MS; MPH, Lab-Incharge (Biochemist), Bangladesh Medical Research Council (BMRC)
Other Study IDs: BBMH/2021/RP-2330
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: HbE Trait; Hemoglobinopathies
Keywords: HbE Disease; Thalassemia; Sickle cell disease
MeSH Terms: conditions — Hemoglobinopathies; Thalassemia; Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention (Diagnostic Test Only): Biochemical Test and detect hemoglobin variants (HPLC, CE)

SUMMARY:
Hemoglobinopathies are inherited disorders that affect haemoglobin and pose a considerable global health challenge. This research addresses the knowledge gap regarding the prevalence of a typical haemoglobin fraction within urban populations by testing the HbA1c test in capillary electrophoresis. Participants will be recruited with careful ethical considerations and informed consent will be obtained. The screening will utilize laboratory techniques to detect abnormal haemoglobin fractions through testing. Statistical methods will be used for data analysis to assess prevalence rates and pinpoint specific haemoglobin variants while considering demographic factors. The project's milestones include planning the study, collecting data (from January 2021 to June 2025), conducting analyses, preparing reports and sharing the findings.

DETAILED DESCRIPTION:
This study is designed as a cross-sectional observational study aimed at detecting and identifying abnormal haemoglobin variants associated with genetic blood disorders, particularly Alpha-thalassemia, Beta-thalassemia, and Sickle Cell Disease, within an urban population. Hemoglobinopathies are among the most prevalent inherited disorders worldwide, yet there remains limited data on their frequency and distribution in metropolitan areas such as Chattogram, Bangladesh, where genetic diversity, lifestyle factors and high population density may influence disease patterns. The rationale behind this study is to provide much-needed baseline epidemiological information that will facilitate early detection, effective prevention strategies and improved clinical management of these conditions.

The primary objective is to identify abnormal haemoglobin types. In contrast, secondary objectives include determining the prevalence of variants, analyzing demographic and lifestyle associations such as age, sex, socioeconomic background and ethnicity and raising community awareness about the importance of genetic carrier screening. The study population will include individuals aged 1 month to seventy years who have been city residents for at least five years and who provide informed consent. Exclusions will apply to individuals requiring emergency care, those already under treatment for known hemoglobinopathies and those unwilling to participate.

The methodology involves stratified random sampling to ensure the study population is representative. Demographic and clinical data such as family history, anaemia, jaundice and history of transfusions will be collected using a structured questionnaire. Venous blood samples (3 mL in EDTA) will be collected from participants and subjected to laboratory investigations. Initial screening will include Complete Blood Count (CBC) and red cell indices such as MCV, MCH and RDW. At the same time, confirmatory testing will be performed using haemoglobin electrophoresis and high-performance liquid chromatography (HPLC) and Capillary Electrophoresis (CE) to quantify and characterize abnormal haemoglobin variants. All results will be entered into a secure, coded database with strict quality control procedures. Statistical analysis will be conducted using SPSS to determine prevalence, distribution and associations between demographic or lifestyle factors.

The expected outcomes include reliable prevalence data of hemoglobinopathies in the selected population, the proportion of carriers versus affected individuals, and correlations with demographic determinants. These findings will guide future diagnostic strategies, inform genetic counselling programs and strengthen targeted public health interventions. Ethical approval will be obtained from the Institutional Review Board and informed consent will be secured from all participants or guardians in the case of minors. Confidentiality will be maintained throughout and individuals with abnormal results will be referred for clinical management and counselling.

Overall, this study will significantly enhance diagnostic awareness, shape health policy and contribute to prevention strategies through community-level interventions. Despite inherent limitations such as its cross-sectional design, potential recall bias in family history reporting and limited access to advanced molecular testing, the study is expected to provide critical insights into the burden of hemoglobinopathies in an urban Bangladeshi population.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the selected metropolitan area.
* All ages (1 Month - 70 Years) and both sexes.
* Willing to provide informed consent.

Exclusion Criteria:

* Refusal to provide informed consent.
* Inaccurate data.

Ages: 1 Month to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comprise individuals residing within the metropolitan area who meet the predefined inclusion criteria. Eligible participants, irrespective of age or sex, will be considered for enrollment, ensuring representation across demographic groups. Participation will be strictly voluntary, and only those who provide informed consent (or assent with parental/guardian consent in the case of minors) will be included in the study. This approach is intended to capture a diverse and representative sample of the target community, thereby enhancing the generalizability and validity of the study findings.
Sampling Method: Non-Probability Sample
Enrollment: 8400 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of abnormal haemoglobin fractions in Chattogram | Day 01, at enrolment
  The proportion of participants identified with abnormal haemoglobin fractions.

SECONDARY OUTCOMES:
Different spectrum of haemoglobin variants | Day 01, on enrolment
  The identification and frequency distribution of specific haemoglobin variants (e.g., HbE, HbS) within the study population.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Science and Technology Chittagong (USTC), Khulshi, Chattogram, Bangladesh

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with other researchers to protect patient confidentiality and comply with institutional and ethical guidelines. Only aggregated, de-identified data may be shared upon reasonable request and with appropriate ethical approvals.